CLINICAL TRIAL: NCT05490264
Title: [68Ga]Ga-NOTA-SNA002 (PD-L1 PET Tracer) for PET/CT in Patients With Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SmartNuclide Biopharma (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SN-2022-01
Record Dates: First submitted 2022-07-08; First posted 2022-08-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumor; Positron-Emission Tomography(PET)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-NOTA-SNA002 (Experimental): A dose of 1mCi-5mCi of [68Ga]Ga-NOTA-SNA002 between 0.1mg to 0.9mg will be administered intravenously over 5minutes in Day 1 of subject enrollment
  Interventions: Biological: [68Ga]Ga-NOTA-SNA002

INTERVENTIONS:
Biological: [68Ga]Ga-NOTA-SNA002 — [68Ga]Ga-NOTA-SNA002（PD-L1 PET Tracer）for Positron Emission Tomography

SUMMARY:
The purpose of this study is to evaluate the safety of [68Ga]Ga-NOTA-SNA002 and investigate the uptake of [68Ga]Ga-NOTA-SNA002 in patients with solid tumors.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be evaluated to determine eligibility for study entry. Patients will receive an injection of [68Ga]Ga-NOTA-SNA002 (1.0-5.0mCi) in Day1 and will undergo PET/CT scanning to determine uptake of [68Ga]Ga-NOTA-SNA002 in tumor lesions and reference tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (including boundary values);
2. Have behavioral ability, and voluntarily participate in this clinical study, and sign the informed consent form (ICF);
3. Performance status (ECOG) score 0-2 points (see Appendix 1 for details);
4. Basal heart rate 60-100 beats/min (including boundary values);
5. Blood pressure measurement < hypertension grade 1 level (including a history of hypertension, systolic blood pressure < 140 and diastolic blood pressure < 90 mmHg by exercise or drug treatment);
6. Patients with confirmed solid tumors;
7. Patients who must have at least one image-measurable lesion according to the evaluation criteria for solid tumors (RECISTv1.1);
8. Imaging results show that at least one tumor lesion can be needle biopsy or surgical treatment to obtain specimens (enhanced CT, enhanced MRI or 18F-FluroDeoxyGlucose(FDG) PET/CT results are acceptable);
9. Patients obtained with immunohistochemical PD-L1 expression results within the previous month.

Exclusion Criteria:

1. Those who are unable to follow this clinical trial protocol well enough to make visits, or undergo relevant examinations, or treatment;
2. Those who have extremely poor nutritional status and cannot tolerate the trial;
3. Known or suspected evidence of active autoimmune disease;
4. Patients taking high doses of hormones, such as more than 20mg of hydrocortisone or 5mg of prednisone in the morning and more than 10mg of hydrocortisone or 2.5mg of prednisone at night；
5. Those with known severe allergy to SNA002, similar drugs or excipients；
6. Patients with brain metastases；
7. Serum virology tests: positive results for any of hepatitis B virus surface antigen, hepatitis C virus antibodies, syphilis-specific antibodies or those who cannot be determined to be negative for human immunodeficiency virus antibodies；
8. Women who are pregnant or breastfeeding.
9. Those who, in the opinion of the investigator, are not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Time of infusion of [68Ga]Ga-NOTA-SNA002 (Day 1) through Visit（Day 6）
  The incident and severity of adverse events per CTCAE V5.0 criteria will be recorded following dose of [68Ga]Ga-NOTA-SNA002.
Changes of vital signs in participants compared with baseline results. | Baseline and 6 hours after infusion of [68Ga]Ga-NOTA-SNA002 (Day 1) and 2 hours after tumor biopsy(Day 2)
  Number of participants in CTCAE 5.0 Stage 1 or higher with vital signs after administration
Changes in laboratory values compared with baseline results. | Baseline and Visit（Day 6）
  Number of participants in CTCAE 5.0 Stage 1 or higher with laboratory examination(e.g. WBC, RBC, HB and other laboratory tests) after administration.
Immunogenicity Analysis of [68Ga]Ga-NOTA-SNA002 | 1 month
  By analyzing anti-SNA002 anti-drug antibody positive rate.
Description of biodistribution patterns of [68Ga]Ga-NOTA-SNA002 on PET | 1 month
  Description of biodistribution patterns of [68Ga]Ga-NOTA-SNA002 on PET.

SECONDARY OUTCOMES:
Standard Uptake Value(max) in tumors | 12 months
  SUVmax quantitative analysis in tumors
Standard Uptake Value(peak) in tumors | 12 months
  SUVpeak quantitative analysis in tumors
Standard Uptake Value(mean) in tumors | 12 months
  SUVmean quantitative analysis in tumors
Correlation of [68Ga]Ga-NOTA-SNA002 uptake in biopsied tumors with PD-L1 measurement by immunohistochemistry (IHC) | 12 months
  Analyze [68Ga]Ga-NOTA-SNA002 uptake in biopsied tumors as determined by SUV-based quantitative measures (SUVmax, SUVpeak, SUVmean) with PD-L1 measurement determined by IHC from biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University; Songbing Qin, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No